CLINICAL TRIAL: NCT02926430
Title: A Randomized, Double-blind, First-in-Human Phase 1 Study to Evaluate the Safety, Tolerability and Immunogenicity of Two Vaccinations of Ad26.RSV.preF One Year Apart in Adults Aged 60 Years and Older in Stable Health
Brief Title: A Study to Evaluate the Safety, Tolerability and Immunogenicity of Two Vaccinations of Ad26.RSV.preF One Year Apart in Adults Aged 60 Years and Older in Stable Health
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Vaccines & Prevention B.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CR108214; VAC18193RSV1003 (Other: Janssen Vaccines & Prevention B.V.)
Record Dates: First submitted 2016-09-22; First posted 2016-10-06 (Estimated); Last update posted 2019-02-19 (Actual); Status verified 2019-02

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

ARMS (5):
- Ad26.RSV.preF 5*10^10 vp (Day 1 and Day 365): Group 1 (Experimental): Participants will receive 5*10^10 viral particles (vp) Ad26.RSV.preF at Day 1 and Day 365 (10 to 13 months after first vaccination).
  Interventions: Biological: Ad26.RSV.preF 5*10^10 vp
- Ad26.RSV.preF 5*10^10 vp (Day 1)- Placebo (Day 365): Group 2 (Experimental): Participants will receive 5*10^10 vp Ad26.RSV.preF at Day 1 and placebo on Day 365 (10 to 13 months after first vaccination).
  Interventions: Biological: Ad26.RSV.preF 5*10^10 vp; Drug: Placebo
- Ad26.RSV.preF 1*10^11 vp (Day 1 and Day 365): Group 3 (Experimental): Participants will receive 1*10^11 vp Ad26.RSV.preF at Day 1 and Day 365 (10 to 13 months after first vaccination).
  Interventions: Biological: Ad26.RSV.preF 1*10^11 vp
- Ad26.RSV.preF 1*10^11 vp (Day 1)- Placebo (Day 365): Group 4 (Experimental): Participants will receive 1*10^11 vp Ad26.RSV.preF at Day 1 and placebo on Day 365 (10 to 13 months after first vaccination).
  Interventions: Biological: Ad26.RSV.preF 1*10^11 vp; Drug: Placebo
- Placebo (Day 1 and Day 365): Group 5 (Experimental): Participants will receive placebo at Day 1 and Day 365 (10 to 13 months after first vaccination).
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: Ad26.RSV.preF 5*10^10 vp — Ad26.RSV.preF will be given at a concentration of 5*10^10 vp/0.5 milliliter (mL).
  Other Names: JNJ-64400141
  Arms: Ad26.RSV.preF 5*10^10 vp (Day 1 and Day 365): Group 1; Ad26.RSV.preF 5*10^10 vp (Day 1)- Placebo (Day 365): Group 2
Biological: Ad26.RSV.preF 1*10^11 vp — Ad26.RSV.preF will be given at a concentration of 1*10^11 vp/0.5 milliliter (mL).
  Other Names: JNJ-64400141
  Arms: Ad26.RSV.preF 1*10^11 vp (Day 1 and Day 365): Group 3; Ad26.RSV.preF 1*10^11 vp (Day 1)- Placebo (Day 365): Group 4
Drug: Placebo — Participants will receive placebo as formulation buffer.
  Arms: Ad26.RSV.preF 1*10^11 vp (Day 1)- Placebo (Day 365): Group 4; Ad26.RSV.preF 5*10^10 vp (Day 1)- Placebo (Day 365): Group 2; Placebo (Day 1 and Day 365): Group 5

SUMMARY:
The purpose of this study is to assess the safety and tolerability of 2 single doses of either 5*10^10 viral particles (vp) or 1*10^11 vp of Ad26.RSV.preF, administered intramuscularly to elderly adults given approximately 12 months apart.

ELIGIBILITY:
Inclusion Criteria:

* Each participant must sign an informed consent form (ICF) indicating that he or she understands the purpose of and procedures required for the study, is willing to participate in the study and attend all scheduled visits, and is willing and able to comply with all study procedures and adhere to the prohibitions and restrictions specified in this protocol
* Before randomization, a woman must be: postmenopausal - A postmenopausal state is defined as no menses for 12 months without an alternative medical cause; and not intending to conceive by any methods
* From the time of first vaccination until 3 months after the first dose of study vaccine, and from the second vaccination through 3 months after, a man who has not had a vasectomy (or if a vasectomy was performed less than 1 year ago and the absence of sperm cannot be verified)
* In the investigator's clinical judgment, participant must be either in good or stable health. Participants may have underlying illnesses such as hypertension, type 2 diabetes, hyperlipoproteinemia, or hypothyroidism, as long as their symptoms/signs are medically controlled. If they are on medication for a condition, the medication dose must have been stable for at least 12 weeks preceding vaccination and expected to remain stable for the duration of the study. Participants will be included on the basis of physical examination, medical history, vital signs, and 12-lead electrocardiogram (ECG) performed at screening
* Participant must be healthy on the basis of clinical laboratory tests performed at screening. If the results of the laboratory screening tests are outside the central laboratory normal reference ranges and additionally within the limits of toxicity Grades 1 or 2 according to the US Food and Drug Administration (FDA) toxicity tables (for tests in the FDA table ), the participant may be included only if the investigator judges the abnormalities or deviations from normal to be not clinically significant and appropriate and reasonable for the population under study. This determination must be recorded in the participant's source documents and initialed by the investigator

Exclusion Criteria:

* Participant has acute illness (this does not include minor illnesses such as diarrhea) or temperature greater than or equal to (>=) 38.0 degree celsius within 24 hours prior to the first dose of study vaccine; enrollment at a later date is permitted
* Participant has a serious chronic disorder, including severe chronic obstructive pulmonary disease or clinically significant congestive heart failure, requirement for supplemental oxygen, end stage renal disease with or without dialysis, clinically unstable cardiac disease, Alzheimer's disease, or has any condition for which, in the opinion of the investigator, participation would not be in the best interest of the participant (for example, compromise well-being) or that could prevent, limit, or confound the protocol-specified assessments
* Participant has had major surgery within the 4 weeks prior to randomization or has planned major surgery through the course of the study
* Participant has chronic active hepatitis B or hepatitis C infection, documented by hepatitis B surface antigen and hepatitis C antibody, respectively
* Participant has human immunodeficiency virus (HIV) type 1 or type 2 infection

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2016-11-08 (Actual); Primary Completion 2018-03-14 (Actual); Study Completion 2019-01-29 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Solicited Local Adverse Events (AEs) for 7 Days After Each Vaccination (Day 1) | 7 days after each vaccination (Day 1)
Number of Participants With Solicited Local Adverse Events (AEs) for 7 Days After Each Vaccination (Day 365) | 7 days after each vaccination (Day 365)
Number of Participants With Solicited Systemic Adverse Events (AEs) for 7 Days After Each Vaccination (Day 1) | 7 days after each vaccination (Day 1)
Number of Participants With Solicited Systemic Adverse Events (AEs) for 7 Days After Each Vaccination (Day 365) | 7 days after each vaccination (Day 365)
Number of Participants With Unsolicited AEs for 28 Days After Each Vaccination | 28 days after each vaccination (from signing the informed consent form [ICF] to Day 29 inclusive)
Number of Participants With Serious Adverse Events (SAEs) Throughout Study | Up to 730 days

SECONDARY OUTCOMES:
Respiratory Syncytial Virus (RSV) Neutralization A2 | Days 1, 29, 183, 365, 393, 547, 730
  Analysis of RSV A2 neutralizing titers of the vaccine-induced immune response will be assessed.
RSV Fusion Protein (F-protein) Enzyme-linked Immunosorbent Assay | Days 1, 29, 183, 365, 393, 547, 730
  Analysis of antibodies binding to RSV F protein in post-fusion and pre-fusion form.
Intracellular Cytokine Staining | Day 1, 29, 183, 365, 393, 547, 730
  The activation of cluster of differentiation 4 (CD4) and cluster of differentiation 8 (CD8) T-cell subsets and their cytokine expression patterns will be determined by flow cytometry after RSV protein peptide stimulation (including, but not limited to CD4/CD8, interleukin [IL-2], interferon gamma [IFN gamma], tumor necrosis factor alpha [TNF-alpha] and/or activation markers, memory, T-helper [cells] Th1/Th2 subtyping).

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Vaccines & Prevention B.V. Clinical Trial, Study Director — Janssen Vaccines & Prevention B.V.
Locations (1):
- Miami, Florida, United States